CLINICAL TRIAL: NCT04261387
Title: A Two-Part (Open-Label Followed by Randomized, Double-Blind, Placebo-Controlled) Phase 1/2 Study to Evaluate the Safety, Tolerability, and Efficacy of Topically Administered LUT014 for the Treatment of Radiation-Induced Dermatitis in Breast Cancer Patients
Brief Title: LUT014 for the Treatment of Radiation Induced Dermatitis in Breast Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lutris Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LUT-RD-02-01
Record Dates: First submitted 2020-02-04; First posted 2020-02-07 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-04

CONDITIONS: Radiation Dermatitis
Keywords: Radiation dermatitis, dermatitis, breast cancer
MeSH Terms: conditions — Radiodermatitis; Dermatitis; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LUT014 Gel (Experimental): LUT014 Gel topical application to the dermatitis area qd for 28 days
  Interventions: Drug: LUT014 Gel
- Placebo for LUT014 Gel (Placebo Comparator)
  Interventions: Drug: Placebo for LUT014 Gel

INTERVENTIONS:
Drug: LUT014 Gel — Topical application qd for 28 days
  Arms: LUT014 Gel
Drug: Placebo for LUT014 Gel — Matching placebo for qd topical application for 28 days
  Arms: Placebo for LUT014 Gel

SUMMARY:
The study will evaluate the safety, tolerability and efficacy of LUT014 gel topically administered in breast cancer patients who developed radiation dermatitis. Subjects enrolled to part 1 will be enrolled to receive the study treatment (open label treatment) for 28 days and will be followed up for 2 months after the completion of study treatment. Subject in Part 2 will be randomized in 1:1 ratio to receive either the study drug or placebo (double-blind treatment) for qd topical application for 28 days and will be followed up for 2 months after the completion of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects diagnosed with stage Tis, T0-T3, N0-N2, M0 Breast Cancer;
2. Subject is ≥18 years at the time of signing the informed consent form (ICF);
3. Radiation dermatitis of Grade 2, based on the NCI CTCAE at the Screening and Baseline (D0) visits;
4. Completed fractionated radiation therapy for breast prior to first dose of study drug (Day 0);
5. A score of ≥ 6 reported in the Dermatology Life Quality Index at the Screening and Baseline Visits;
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
7. Females of child-bearing potential must have a negative pregnancy test at screening and must agree to use an effective contraception method* or abstain from sex throughout the study until Day 83;
8. Expected life expectancy greater than 6 months

Exclusion Criteria:

1. Bilateral breast irradiation;
2. Planned internal mammary node irradiation with electrons. Planned photon coverage of internal mammary chain nodes is acceptable for inclusion in this study;
3. Planned partial breast accelerated irradiation;
4. Any cutaneous infection or significant skin disease at Screening or Baseline (Day 0) other than the dermatitis in the area(s) irradiated during fractionated radiation therapy;
5. T4 breast cancer or direct skin involvement by breast cancer;
6. Breast implants or underwent breast reconstruction;
7. Any cancer other than breast cancer within 3 years of Screening, except for carcinoma in situ of the cervix;
8. Pregnant or lactating;
9. History of active systemic lupus erythematosus or scleroderma that is believed to increase the risk of developing radiation-induced dermatitis or its severity;
10. Clinically significant co-morbid diseases
11. Treatment with a serine/threonine-protein kinase B-Raf (B-Raf) inhibitor, including but not limited to Zelboraf® (vemurafenib), Tafinlar® (dabrafenib), Braftovi® (encorafenib), and Nexavar® (sorafenib), within 30 days or 5 half-lives of the drug prior to Screening, whichever is longer;
12. Treatment with a topical corticosteroid o the irradiated chest area within 14 days prior to Baseline (Day 0).
13. Treatment with a systemic corticosteroid within 14 days prior to Baseline (Day 0), except for low dose systemic corticosteroids (e.g., 8-20 mg dexamethasone or comparable) given for up to one or two days every two weeks as part of standard of care for the prevention or treatment of chemotherapy-induced nausea and vomiting (CINV);
14. Treatment with any investigational drug within 30 days or 5 half-lives of drug prior to Screening, whichever is longer;
15. Known hypersensitivity to any of the inactive ingredients of the study drug.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-01-30 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE (Part 1 subjects) | 12 weeks (83 days)
  Common Terminology Criteria for Adverse Events Version 5.0
Change in the severity of radiation dermatitis based on self reporting Dermatology QoL questionnaire (Part 2 subjects) | 14 Days
  Dermatology Life Quality Index questionnaire

SECONDARY OUTCOMES:
Change in the severity of radiation dermatitis assessed by CTCAE (Part 1 subjects) | 12 weeks (83 days)
  CTCAE grading scale for dermatitis radiation
Change in the severity of radiation dermatitis assessed by RTOG/EORTC (part 1 subjects) | 12 weeks (83 days)
  Toxicity criteria of the Radiation Therapy Oncology Group (RTOG) and the European Organization for Research and Treatment of Cancer (EORTC)
Change in the severity of radiation dermatitis based on self reporting Dermatology QoL questionnaire | 12 weeks (83 days)
  Dermatology Life Quality Index questionnaire (part 1 subjects)
Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE (Part 2 subjects) | 12 weeks (83 days)
  CTCAE grading scale for dermatitis radiation

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Columbus Regional Research Institute, Llc, Columbus, Georgia
  - Willis-Knighton Cancer Center, Shreveport, Louisiana